CLINICAL TRIAL: NCT06120699
Title: Effectiveness of Pelvic Floor Muscle Training Including 360 Degree Expanded Diaphragm Exercises in Women With Stress Urinary Incontinence: Double-Blind Randomized Controlled Study
Brief Title: 360 Degree Expanded Diaphragm Exercises in Women With Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Assistant Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYY_İEÜ_2
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Stress Urinary Incontinence; Diaphragmatic Breathing; Pelvic Floor Muscle Exercise; Intra-abdominal Pressure
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: This is a prospective double-blind randomized controlled study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 360 Degree Expanded Diaphragm Exercises (Experimental): Volunteers who complain of urinary incontinence in situations such as coughing, sneezing and laughing, who have been diagnosed with stress or stress-predominant mixed urinary incontinence by a Gynecology and Obstetrics physician, and who meet the inclusion criteria will be included in the study.
  Interventions: Other: Pelvic floor muscle training with 360 degree expanded diaphragm exercises
- Standard Diaphragm Exercises (Active Comparator): Volunteers who complain of urinary incontinence in situations such as coughing, sneezing and laughing, who have been diagnosed with stress or stress-predominant mixed urinary incontinence by a Gynecology and Obstetrics physician, and who meet the inclusion criteria will be included in the study.
  Interventions: Other: Pelvic floor muscle training with standard diaphragm exercises

INTERVENTIONS:
Other: Pelvic floor muscle training with 360 degree expanded diaphragm exercises — Women in this group will be taught 360-degree expanded diaphragm exercises with the Ohmbelt device. Two Ohmbelt devices will be used in this study. The anterior sensor will be placed in the inguinal cavity to visualize the expansion of the anterior abdominal wall, and the posterior sensor will be placed contralaterally in the upper lumbar triangle to visualize the expansion of the posterior wall. The protocol of breathing exercises is inspiration and expiration time of 6 seconds, 10 repetitions and 3 sets. Pelvic floor muscle training will be given with the NeuroTract Myoplus 4 PRO EMG biofeedback device. The training protocol: Each patient will be asked to contract close to the maximum pelvic floor muscle contraction for slow muscle contraction, maintain the contraction for 6-8 seconds, and then perform fast muscle contractions 3-4 times. This cycle is 1 set, 8-12 repetitions. A total of 3 sets will be applied.
  Arms: 360 Degree Expanded Diaphragm Exercises
Other: Pelvic floor muscle training with standard diaphragm exercises — Women in this group will be taught standard diaphragm exercises. In the supine position, with the head and knees supported by a pillow, the patient will first be asked to close his or her eyes to focus. With one hand on the chest and the other hand on the abdomen, "Take a deep breath through your nose and direct all the air as much as possible under your lower hand. inflate your belly. Now exhale all the air slowly through your mouth." The protocol of breathing exercises is inspiration and expiration time of 6 seconds, 10 repetitions and 3 sets. Pelvic floor muscle training will be given with the NeuroTract Myoplus 4 PRO EMG biofeedback device. The training protocol: Each patient will be asked to contract close to the maximum pelvic floor muscle contraction for slow muscle contraction, maintain the contraction for 6-8 seconds, and then perform fast muscle contractions 3-4 times. This cycle is 1 set, 8-12 repetitions. A total of 3 sets will be applied.
  Arms: Standard Diaphragm Exercises

SUMMARY:
This study was planned to examine and compare the effects of standard diaphragm exercises with Pelvic floor muscle exercises (PFME) and 360-degree expanded diaphragm exercises with PFME on urinary symptoms, PFM functions and quality of life in women with stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman,
* Participating in the research voluntarily,
* Being between the ages of 18-62,
* Ability to read and write Turkish,
* Not having any mental problems that would prevent cooperation and understanding,
* Having a complaint of stress urinary incontinence or stress-predominant mixed urinary incontinence.

Exclusion Criteria:

* Having received pelvic floor training before,
* Having a neurological disease,
* Pelvic organ prolapse stage is stage 2 or higher,
* Having fecal incontinence,
* Being pregnant,
* Lower extremity problems that may affect the pelvic structure (conditions such as lower extremity inequality, total hip arthroplasty)
* Having an active lower urinary tract infection,
* Having respiratory system diseases such as chronic obstructive pulmonary disease and asthma,
* Having undergone hysterectomy surgery.

Ages: 18 Years to 62 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Change of Pelvic floor muscle contraction during Valsalva | at baseline, at 8th week
  Pelvic floor muscle contraction during Valsalva will be evaluated with the NeuroTract Myoplus 4 PRO EMG device. A disposable, cylindrical endovaginal probe will be used to record pelvic floor muscle electromyographic activity. The evaluation will be carried out as stated in previous studies, and the women are told: "Take as deep a breath as possible, pinch your nose with your thumb and index finger and close your mouth, try to breathe out against the now closed respiratory system." instructions will be given. For a clearer understanding, the expression "pretend to strain" will also be used. The probe will be manually supported by the investigator throughout the testing procedure to prevent the pressure probe from moving and losing contact with the PTK during evaluation. 2 seconds of reflex PFM activity will be recorded in μV.

SECONDARY OUTCOMES:
Change of urinary symptoms | at baseline, at 8th week
  The severity of women's incontinence will be questioned with the Incontinence Severity Index.
Change of quality of life score | at baseline, at 8th week
  Urinary incontinence symptoms and their impact on quality of life will be evaluated with the International Urinary Incontinence Questionnaire Form.
Change of Pelvic floor muscle maximum voluntary contraction | at baseline, at 8th week
  Maximum voluntary contraction of women will be evaluated with the NeuroTract Myoplus 4 PRO EMG device. A disposable, cylindrical endovaginal probe will be used to record pelvic floor muscle electromyographic activity. MVC, average peak activation results during three PFM contractions will be expressed in μV and percentage (%).
Change of maximum inspiratory pressure | at baseline, at 8th week
  A non-invasive, RP Check brand electronic pressure measuring device (MD Diagnostics Ltd., Maidstone, UK) will be used to measure maximum inspiratory pressure.
Change of maximum expiratory pressure | at baseline, at 8th week
  A non-invasive, RP Check brand electronic pressure measuring device (MD Diagnostics Ltd., Maidstone, UK) will be used to measure maximum expiratory pressure.
Subjective perception of improvement | at 8th week
  Women's subjective perception of improvement was assessed using the Global Perception of Improvement scale
Change of Social Activity Participation | at baseline, at 8th week
  The Social Activity Index will be used, in which nine social situations are selected to represent situations in which women have problems in social participation due to urinary incontinence.
Change of average number of urinary incontinence | at baseline, at 8th week
  Women will be asked to complete a bladder diary reflecting the daily activity patterns of the bladder for 3 consecutive days.
Change of Pelvic floor muscle strength | at baseline, at 8th week
  Vaginal palpation method will be used to measure pelvic floor muscle strength. (Modified Oxford Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yakıt Yeşilyurt, PhD, Principal Investigator — Izmir University of Economics
Locations (1):
- Izmir University of Economics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No